CLINICAL TRIAL: NCT06071533
Title: Effectiveness and Safety of Danshen Injection for Acute Kidney Injury in Primary Nephrotic Syndrome
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Tianxin Chen, associate chief physician, First Affiliated Hospital of Wenzhou Medical University
Other Study IDs: KY2023-R157
Record Dates: First submitted 2023-09-27; First posted 2023-10-06 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Acute Kidney Injury; Nephrotic Syndrome; Nephropathy
Keywords: acute kidney injury; nephrotic syndrome; Danshen injection
MeSH Terms: conditions — Acute Kidney Injury; Nephrotic Syndrome; Kidney Diseases | interventions — Dandshen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Danshen Injection(DS group): patients received Danshen Injection
  Interventions: Drug: Dandshen
- Sportive Care group (SC group): patients received sportive care without Danshen Injection

INTERVENTIONS:
Drug: Dandshen — Dandshen injection 20ml /day
  Groups: Danshen Injection(DS group)

SUMMARY:
The goal of this real-world observational study is to evaluate the effectiveness and safety of the Chinese herbal-derived therapeutic Danshen injection following immunosuppressive therapy and prophylactic anticoagulation with low molecular heparin for acute kidney injury in primary nephrotic syndrome. The main questions to answer are:

Whether or not Danshen injection is beneficial for acute kidney injury patients in primary nephrotic syndrome patients.

Whether or not Danshen injection will increase the bleeding risk in primary nephrotic syndrome patients receiving low molecular heparin.

Participants' information will be retrieved from hospital files stored in medical records and the electronic patient data registry. Participants received Danshen injection will be compared with control group to evaluate the recovery of renal function and side effects.

DETAILED DESCRIPTION:
Background and objectives： Acute kidney injury (AKI) is a common complication of primary nephrotic syndrome (PNS), affecting approximately 23.7% to 34% of PNS patients. No randomized clinical trials and clinical drug intervention studies focus on renal function recovery of AKI in PNS patients. The aim of this study is to assess the clinical effectiveness and safety of a common traditional Chinese herbal medicine (Danshen) in PNS with AKI patients.

Methods:

This study will be a retrospective cohort study of PNS with AKI patients. Renal function recovery and adverse events of the patients receiving Danshen injection(DS group) will be compared with that of the patients with supportive care(SC group) .The study will be conducted using Hospital Information System of the First Affiliated Hospital of Wenzhou Medical University which has longitudinal health information on over 6 million predominantly privately insured individuals and includes over 50 million followup records. The data of inpatients diagnosed with nephrotic syndrome will be reviewed retrospectively. Patients' information includes socio-demographic characteristics, administrative claims (diagnosis and procedure codes), medical histories, laboratory test results and pharmacy claims. PNS wih AKI inpatients will be enrolled. The baseline characteristics will be propensity-score matched. The outcomes are complete and partial renal function recovery for effectiveness analysis and severe bleeding events for safety analysis. Comparisons of cumulative recovery rate will be performed by Kaplan-Meier curves and log-rank test. Risks for outcomes will be assessed using Cox proportional hazard regression models.

ELIGIBILITY:
Inclusion Criteria:

1. age >=20yr;
2. Patients must have at least one "Evaluation and Management"visit with a diagnosis of PNS 6 months before index date;
3. Patients must have AKI at the index date.

Exclusion Criteria:

1. Secondary necrotic syndrome, which is define as necrotic syndrome caused by diabetic nephropathy, lupus nephritis, castleman syndrome, cryoglobulinemia, lymphoma, systemic vasculitis, hepatitis C associated nephritis, hepatitis B associated nephritis, monoclonal immunoglobulinemia, amyloidosis, Sjogren's disease, myeloma, macroglobulinemia and Henoch-Schonlein purpura nephritis；
2. Cancer patients；
3. Liver cirrhosis；
4. Transplant patients;
5. Guillain-Barre syndrome；
6. Maintain Remission in PNS；
7. Chronic renal failure；
8. PNS without AKI;
9. PNS with autosomal dominant polycystic kidney disease;
10. AKI caused by bleeding, haemolytic uraemic syndrome, malignant hypertension，IgG4 related tubulointerstitial nephritis, infection, acute coronary syndrome or heart failure, obstructive nephropathy and nephrotoxic drug ;
11. PNS accompanied with pulmonary embolism, acute cerebrovascular accident,Pregnancy;
12. Acute rapid progressive or Crescentic Glomerulonephritis;
13. Patients without valid data .

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted using Hospital Information System of the First Affiliated Hospital of Wenzhou Medical University which has longitudinal health information on over 6 million predominantly privately insured individuals and includes over 50 million followup records. 3873 patients with nephrotic syndrome will be reviewed retrospectively. Patients' information includes socio-demographic characteristics, administrative claims (diagnosis and procedure codes), medical histories, laboratory test results and pharmacy claims.
Sampling Method: Non-Probability Sample
Enrollment: 441 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
complete renal function recovery renal function recovery recovered to normal level | 6 months
  renal function recovery recovered to normal level
partial renal function recovery | 6 months
  Scr has a 30% or greater reduction from peak values,but not to normal level

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen T, Zhou Y, Chen X, Chen B, Pan J. Acute kidney injury in idiopathic membranous nephropathy with nephrotic syndrome. Ren Fail. 2021 Dec;43(1):1004-1011. doi: 10.1080/0886022X.2021.1942913. PMID 34157952
- [Background] Lu H, Xiao L, Song M, Liu X, Wang F. Acute kidney injury in patients with primary nephrotic syndrome: influencing factors and coping strategies. BMC Nephrol. 2022 Mar 5;23(1):90. doi: 10.1186/s12882-022-02720-y. PMID 35247980
- [Background] Chen T, Lv Y, Lin F, Zhu J. Acute kidney injury in adult idiopathic nephrotic syndrome. Ren Fail. 2011;33(2):144-9. doi: 10.3109/0886022X.2011.553301. PMID 21332335
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Glomerular Diseases Work Group. KDIGO 2021 Clinical Practice Guideline for the Management of Glomerular Diseases. Kidney Int. 2021 Oct;100(4S):S1-S276. doi: 10.1016/j.kint.2021.05.021. No abstract available. PMID 34556256
- [Background] Lian F, Wu L, Tian J, Jin M, Zhou S, Zhao M, Wei L, Zheng Y, Wang Y, Zhang M, Qin W, Wu Z, Yuan CS, Tong X. The effectiveness and safety of a danshen-containing Chinese herbal medicine for diabetic retinopathy: a randomized, double-blind, placebo-controlled multicenter clinical trial. J Ethnopharmacol. 2015 Apr 22;164:71-7. doi: 10.1016/j.jep.2015.01.048. Epub 2015 Feb 7. PMID 25666427
- [Background] Lyu J, Xue M, Li J, Lyu W, Wen Z, Yao P, Li J, Zhang Y, Gong Y, Xie Y, Chen K, Wang L, Chai Y. Clinical effectiveness and safety of salvia miltiorrhiza depside salt combined with aspirin in patients with stable angina pectoris: A multicenter, pragmatic, randomized controlled trial. Phytomedicine. 2021 Jan;81:153419. doi: 10.1016/j.phymed.2020.153419. Epub 2020 Dec 10. PMID 33360345
- [Background] Zhang Y, Xie Y, Liao X, Jia Q, Chai Y. A Chinese patent medicine Salvia miltiorrhiza depside salts for infusion combined with conventional treatment for patients with angina pectoris: A systematic review and meta-analysis of randomized controlled trials. Phytomedicine. 2017 Feb 15;25:100-117. doi: 10.1016/j.phymed.2017.01.002. Epub 2017 Jan 6. PMID 28190464
- [Background] Lameire NH, Levin A, Kellum JA, Cheung M, Jadoul M, Winkelmayer WC, Stevens PE; Conference Participants. Harmonizing acute and chronic kidney disease definition and classification: report of a Kidney Disease: Improving Global Outcomes (KDIGO) Consensus Conference. Kidney Int. 2021 Sep;100(3):516-526. doi: 10.1016/j.kint.2021.06.028. Epub 2021 Jul 9. PMID 34252450
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Result] Menon S. Acute Kidney Injury in Nephrotic Syndrome. Front Pediatr. 2019 Jan 14;6:428. doi: 10.3389/fped.2018.00428. eCollection 2018. PMID 30693275